CLINICAL TRIAL: NCT02647931
Title: Muscle Tension Dysphagia Treatment Efficacy
Brief Title: The Role of Therapy for Muscle Tension Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David G. Lott, M.D., Physician, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-006933
Record Dates: First submitted 2015-11-13; First posted 2016-01-06 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Muscle Tension Dysphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Voice Therapy for Muscle Tension Dysphagia (Experimental): Voice therapy for Muscle Tension Dysphagia patients.
  Interventions: Behavioral: Voice therapy for Muscle Tension Dysphagia

INTERVENTIONS:
Behavioral: Voice therapy for Muscle Tension Dysphagia — Voice therapy for Muscle Tension Dysphagia

SUMMARY:
Muscle tension dysphagia is a novel diagnostic taxonomy describing a subset of patient population with reported dysphagia who exhibit normal oropharyngeal and esophageal swallowing function as evidenced by videofluoroscopic swallow study. These patients also demonstrate abnormal supraglottic muscle tension during laryngoscopy as well as signs of laryngeal hypersensitivity and laryngopharyngeal reflux. Treatment of these patients with Proton Pump Inhibitor (PPI) therapy is a common practice however voice therapy invention targeting the unloading of the supraglottic muscle tension has been shown to be highly effective in symptom resolution per the investigators' clinical experience. The study is designed to answer efficacy of treatment being offered to patients with muscle tension dysphagia.

ELIGIBILITY:
Inclusion Criteria

* Age 18-99
* Diagnosed with Muscle Tension Dysphagia

Exclusion Criteria

* Physical or emotional disorder preventing the completion of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-11; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Improvement of dysphagia measured via patient self-report measures | Duration of therapy, approximately 2 months
  Number of participants who report improvement of dysphagia symptoms following therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kang, CCC-SLP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States